CLINICAL TRIAL: NCT04789668
Title: Phase I/II Trial of BINTRAFUSP ALFA (M7824) and Pimasertib for Treatment of Intracranial Metastases
Brief Title: Bintrafusp Alfa and Pimasertib for the Treatment of Patients With Brain Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1091; NCI-2021-00219 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1091 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-08; First posted 2021-03-09 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Hematopoietic and Lymphoid Cell Neoplasm; Hormone Receptor Positive Breast Adenocarcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Triple-Negative Breast Carcinoma; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Hematologic Neoplasms; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Neoplasm Metastasis; Melanoma; Triple Negative Breast Neoplasms; Lung Neoplasms | interventions — bintrafusp alfa protein, human; N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (bintrafusp alfa, pimasertib) (Experimental): Patients receive bintrafusp alfa IV over 1 hour every 2 weeks and pimasertib PO BID on days 1-28. Treatment repeats every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bintrafusp Alfa; Drug: Pimasertib; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Bintrafusp Alfa — Given IV
  Other Names: Anti-PDL1/TGFb Trap MSB0011359C; M7824; MSB0011359C
Drug: Pimasertib — Given PO
  Other Names: AS703026; EMD 1036239; MSC1936369
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase I/II trial studies the best dose and effect of pimasertib in combination with bintrafusp alfa in treating patients with cancer that has spread to the brain (brain metastases). Immunotherapy with bintrafusp alfa, a bifunctional fusion protein composed of the monoclonal antibody anti-PD-L1 and TGF-beta, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Pimasertib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving pimasertib and bintrafusp alfa may help to prevent or delay the cancer from progressing (getting worse) and/or coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish safety profile and recommended phase II dose for combining pimasertib with bintrafusp alfa (M7824) in patients with brain metastases. (Phase I)

II. Time to intracranial progression (defined as progression of existing lesions and development of new lesions by modified Response Evaluation Criteria in Solid Tumors [RECIST] 1.1). (Phase II)

III. Overall survival. (Phase II)

SECONDARY OBJECTIVES:

I. Intracranial progression 6, 12 and 18 months.

II. Intracranial objective response rate as measured by Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM), immunotherapy (i)RANO, and RECIST 1.1.

III. Time to second intracranial progression after salvage stereotactic radiosurgery (SRS).

IV. Overall survival rate at 6, 12 and 18 months.

V. Frequency of grade 3+ intracranial toxicities at 4 weeks, and 3, 6, 9, 12 and 18 months.

VI. Frequency of extracranial progression and response rate at 8 weeks, and 3, 6, 9, 12 and 18 months.

VII. Frequency of neurocognitive decline at 6, 12 and 18 months (optional).

VIII. Changes in neurocognitive function and health-related quality of life.

IX. Dose, duration and frequency of steroid use for symptomatic management.

EXPLORATORY OBJECTIVES:

I. Identify molecular and/or immunological markers from biospecimens (tissue, blood, and cerebrospinal fluid [CSF]) that are associated with treatment response and toxicity.

II. Identify imaging biomarkers of response and toxicity (acute radiation effect/radionecrosis and neurocognitive changes) from multiparametric magnetic resonance imaging (MRI) and/or delayed positron emission tomography (PET) that predict treatment response and toxicity.

III. Identify correlative or surrogative relationship between systemic (blood) and imaging markers and treatment outcomes.

OUTLINE: This is a phase I, dose-escalation study of followed by a phase II dose-expansion study.

Patients receive bintrafusp alfa intravenously (IV) over 1 hour every 2 weeks and pimasertib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, every 6 weeks during year 1, and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Life expectancy > 12 weeks
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* At least one measurable untreated brain lesion >= 0.5 cm and < 3.0 cm in the longest axis according to modified RECIST 1.1
* Prior stereotactic radiosurgery (SRS) with up to 3 lesions treated with at least a 14 day interval is allowed as long as the previous treatment volume does not overlap with the current targets
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Subjects must be free of neurologic signs and symptoms related to metastatic brain lesions and must not have required or received systemic corticosteroid therapy in the 10 days prior to beginning protocol therapy
* Prior treatment with immunotherapy and targeted therapy allowed as long as it did not include a combination of MEK inhibitor (i) + anti-PD(L)-1 antibody and is > 14 days prior to start of protocol therapy. All tumor types will be eligible and included in the dose escalation phase. Dose expansions will include 10 patients each from lung, breast, and melanoma
* Patients with melanoma must have received prior PD-1 based therapy and have evidence of progression
* Patients with non-small cell lung cancer (NSCLC) must have received prior PD-1 based therapy and have evidence of progression
* Patients with triple-negative breast cancer (TNBC) and hormone receptor positive (HR+) are included (any number of prior lines of therapy-including immuno-oncology [IO] naive patients)
* For HR+ patients, patients are allowed to receive endocrine therapy with or without CDK4/6 inhibitors per treating physician discretion (Arimidex, letrozole, exemestane, or fulvestrant)
* Systematic radiation therapy is allowed (> 14 day washout)
* Prior platinum-based chemotherapy for NSCLC patients is allowed
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelets >= 100 000/uL
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for participant with creatinine levels > 1.5 x institutional ULN

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Women of child-bearing potential (WOCBP) must not be breastfeeding and must have a negative pregnancy test within 3 days prior to initiation of dosing. She must agree to use an acceptable method of birth control from the time of the negative pregnancy test up to 120 days after the last dose of study drug. WOCBP must agree to adhere to the contraceptive guidance

  * Note: A female participant is eligible to participate if she is not a woman of childbearing potential
* Fertile men must agree to use an acceptable method of birth control while on study drug and up to 120 days after the last dose of study drug and also refrain from donating sperm during this period
* All associated toxicity from previous or concurrent cancer therapy must be resolved (to =< grade 1 or baseline) prior to study treatment administration. Steroids for physiological replacement are allowed

Exclusion Criteria:

* Patients with clinical or radiographic evidence of leptomeningeal disease
* Those who experienced grade 3 or 4 neurotoxicity from prior SRS
* Prior external beam radiation to the brain or whole brain radiation
* Contraindications to MRI (implanted metal device or foreign bodies) or MRI contrast (insufficient renal function or allergy)
* Subjects with major medical, neurologic or psychiatric condition who are judged as unable to fully comply with study therapy or assessments should not be enrolled
* Active secondary malignancy unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the principle investigator (PI). Examples of the latter include basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, and isolated elevation of prostate-specific antigen. Subjects with a completely treated prior malignancy and no evidence of disease for >= 2 years are eligible
* Has a known history of or is positive for hepatitis B (hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus infection (note treated and cured history of hepatitis C is allowed) (hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)

  * Note: Without known history, testing needs to be performed to determine eligibility. Hepatitis C antibody (Ab) testing is allowed for screening purposes in countries where HCV RNA is not part of standard of care
* Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority
* The use of corticosteroids is not allowed for 10 days prior to initiation of therapy (based upon 5 times the expected half-life of dexamethasone) except patients who are taking steroids for physiological replacement. If alternative corticosteroid therapy has been used, consultation with the PI is required to determine the washout period prior to initiating study treatment
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study initiation. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Major surgical procedure, open biopsy (excluding skin cancer resection), or significant traumatic injury within 14 days of initiating study drug (unless the wound has healed) or anticipation of the need for major surgery during the study
* Non-healing wound, ulcer, or bone fracture
* Women who are breast-feeding or pregnant
* Subjects with a history of serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, bleeding diathesis or recent major bleeding events or other illness considered by the Investigator as high risk for investigational drug treatment
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than 1 month before the start of study medication)
* History of clinically significant cardiac disease or congestive heart failure > New York Heart Association (NYHA) class 2. Subjects must not have unstable angina (anginal symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months
* Investigational drug use within 14 days (or 5 half-lives, whichever is longer) of the first dose of bintrafusp alfa and/or pimasertib
* Has a history of (grade 3 or 4) non-infectious pneumonitis that required steroids or current pneumonitis
* Retinal degenerative disease (hereditary retinal degeneration or age-related macular degeneration), history of retinal vein occlusion (RVO) or any eye condition that would be considered as risk factor for RVO (e.g. uncontrolled glaucoma or ocular hypertension)
* Creatine phosphokinase level at baseline National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 (> 2.5 x ULN - 5 x ULN) and/or previous history of myositis or rhabdomyolysis
* For NSCLC cohort patients whose tumor exhibit activating EGFR mutation, ALK or ROS translocation and have a standard of care molecular targeted therapy available for these mutations, will be excluded from this study. Patients who progressed or could not tolerate these standard of care molecular targeted agents are eligible for this study. Lung adenocarcinoma patients may be consented prior to the EGFR and ALK status being known, but EGFR and ALK status must be determined prior to initiating therapy
* Administration of live, attenuated vaccine therapies for the prevention of infectious diseases within 4 weeks prior to day 1 of treatment and during therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate | Up to 2 years
Incidence of intracranial and extracranial toxicities and dose-limiting toxicities (Phase I) | Up to 90 days
  Will be summarized by grade, relationship, time during the treatment, etc., for each dose in each group.
Recommended phase II dose (Phase I) | At 4 weeks after first administration of treatment
  The recommended phase II dose is defined as the highest dose level with no more than 1 patient with dose-limiting toxicity out of 6 patients that are treated.
Time to intracranial progression (Phase II) | From the time of study enrollment to intracranial progression (event) or the last follow-up date if the patient has not developed the intracranial progression yet, assessed up to 2 years
  Will be determined by modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and estimated using Kaplan-Meier method with 95% confidence interval.
Overall survival (Phase II) | From treatment start date to death, assessed up to 2 years
  Will be estimated using Kaplan-Meier method, both with 95% confidence interval.

SECONDARY OUTCOMES:
Intracranial progression | From the time of study enrollment to intracranial progression (event) or the last follow-up date if the patient has not developed the intracranial progression yet, assessed up to 18 months
  Will be determined by modified RECIST 1.1 and estimated and reported with 95% confidence interval utilizing the method of Kaplan and Meier. Will be performed overall and within each treatment group. Completing risk analysis may be considered by treating events outside of intracranial disease progression (e.g. events such as extracranial disease progression, early dropout due to toxicity, or death) as competing risks.
Time to extracranial progression | From the time of study enrollment to extracranial progression (event) or thelast follow-up date if the patient has not developed the extracranial progression yet, assessed up to 18 months
  Will be determined by modified RECIST 1.1. The cumulative incidence rate may be estimated by competing risk analysis treating events outside of extracranial disease progression (e.g. events such as intracranial disease progression, early dropout due to toxicity, or death) as competing risks.
Best achieved extracranial objective response rate | Up to 2 years
  Will be reported for each patient. The frequency of extracranial objective response will be reported overall and within each treatment group.
Duration of response | From date of first imaging identifying partial response (PR) or complete response (CR) until the date of first imaging identifying progressive disease is noted, assessed up to 2 years
  Will be assessed in patients who achieve extracranial, PR or CR via RECIST 1.1 criteria and calculated utilizing the Kaplan-Meier method with reporting of the median and range overall and within each treatment group.
Dose, duration and frequency of steroid use for symptomatic management | Up to 2 years
  Will record and report steroid requirements for symptom management overall and within each treatment group. Patients who require at least 4 mg of dexamethasone/day for symptom management will be considered as requiring high dose steroids.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein A Tawbi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT04789668/Prot_SAP_000.pdf